CLINICAL TRIAL: NCT02050997
Title: Identification of Predictive Plasma Biomarkers in Pancreatic Ductal Adenocarcinoma (PDAC Plasma Biomarker Study)
Brief Title: Plasma Biomarkers P-DAC, V1
Status: Terminated | Type: Observational
Why Stopped: As per the HRBs new funding model, HRBs investment will not support costs associated with routine patient care or translational studies, biobanks, patient registries and questionnaires. Therefore, a decision was made to cease further study follow up.
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: CTRIAL-IE (ICORG) 12-31
Record Dates: First submitted 2014-01-24; First posted 2014-01-31 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- B: Unresectable or metastatic PDAC patients who will receive standard treatment of CT +/- radiotherapy
- A: Resectable PDAC patients who will receive standard treatment of CT +/- radiotherapy

SUMMARY:
This is an exploratory, translational, non-interventional and multi-centre clinical study. The aim of the study is to identify predictive plasma biomarkers of response to chemotherapy in PDAC.

DETAILED DESCRIPTION:
This study will involve two cohort groups, all patients involved will have PDAC.

Cohort A: Target is 80 resectable PDAC patients who will receive standard treatment of chemotherapy +/- radiotherapy

Cohort B:

* Cohort B1 = Target is 80 unresectable locally advanced PDAC patients who will receive standard treatment of chemotherapy +/- radiotherapy.
* Cohort B2 = Target is metastatic PDAC patients who will receive standard treatment of chemotherapy +/- radiotherapy.

Control patients: Target is 50, with acute pancreatitis admitted to hospital for observation/treatment.

Blood samples will be taken at the following time points:

* prior to resection, whenever feasible for cohort A
* prior to CT, for both cohort A and B
* during CT, for both cohort A and B
* follow-up, approximately every 3 to 6 months for two years for cohort A

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Ability to give written informed consent
* Histologically or cytologically-confirmed PDAC
* Patients who will receive standard treatment of CT +/- radiotherapy and present with:

Cohort A: resectable cancer OR Cohort B.1: unresectable locally advanced cancer OR Cohort B.2: metastatic cancer

* Eastern Cooperative Oncology Group (ECOG) Performance status 0 - 2

Exclusion Criteria:

* Presence of medical or psychiatric conditions, which, in the opinion of the investigator, would potentially pose a risk to the patient in participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients on this study must have pancreatic ductal adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2014-05-26 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Time to disease recurrence | Blood samples analysed up to 2 year follow up, estimated 4 years in total
  Identify plasma biomarkers that are predictive for response to treatment as defined by time to recurrence

SECONDARY OUTCOMES:
Rate of progression free survival | Blood samples analysed up to 2 year follow up, estimated 4 years in total
  To discover plasma biomarkers that are predictive for response to treatment as defined by progression free survival
Accuracy, sensitivity, specificity and concordance index | For the duration of study, expected 4 years
  Aim to validate a panel of predictive plasma biomarkers proving its accuracy, sensitivity, specificity and to investigate their expression at tissue level gaining a further understanding of cancer and/or host related proteins in disease response and progression

CONTACTS AND LOCATIONS:
Locations (9):
- Ireland (9):
  - Beacon Hospital, Dublin, Dublin 18
  - Our Lady of Lourdes Hospital Drogheda, Drogheda, Louth
  - Bon Secours, Cork
  - Beaumont Hospital, Dublin
  - St Vincent's Hospital, Dublin
  - Galway University Hospital, Galway
  - Midwestern Regional Hospital, Limerick
  - Adelaide Meath National Childrens Hospital, Tallaght
  - Waterford Regional Hospital, Waterford